CLINICAL TRIAL: NCT00002173
Title: An Expanded Access Open Label Protocol of Remune (HIV-1 Immunogen) in HIV-1-Infected Adults With CD4 Count 550 Cells /Ml and Greater.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Immune Response Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 094; 902
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-06

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS Vaccines; CD4 Lymphocyte Count; Salk HIV Immunogen
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — HIV-1 immunogen, incomplete Freund's adjuvant

INTERVENTIONS:
Biological: HIV-1 Immunogen

SUMMARY:
To provide an alternative therapy to HIV-infected patients for whom there is no comparable or satisfactory alternative drug or therapy available.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositivity.
* CD4 counts >= 550 cells/ml.

NOTE:

* If a patient's CD4 count is 550 to 600 cells/ml, the patient must either rescreen within 30 days for Study 806 or wait 6 months before entering the expanded access program.
* Patient must have failed or been intolerant to other comparable or alternative marketed therapies or must not be a candidate for such therapies.
* Patient must not meet inclusion criteria for other Remune trials.
* Patient must have laboratory tests within specified limits.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Clinically significant cardiac, hepatic, renal or gastrointestinal dysfunction.
* Current participation in a Remune study.

Concurrent Medication:

Excluded:

* Use of any immune-modulating drugs.
* Induction therapy or initiation of new treatment regimen for an AIDS-defining condition.
* Current participation in a Remune study.

Patients with any of the following prior conditions are excluded:

Previous participation in a Remune study.

Prior Medication:

Excluded:

* Previous participation in a Remune study.

Excluded within 30 days of study entry:

* Use of any immune-modulating drugs.
* Induction therapy or initiation of new treatment regimen for an AIDS-defining condition within 30 days of Day 1 visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Immune Response Corp, Carlsbad, California, United States